CLINICAL TRIAL: NCT06439147
Title: U-shaped vs T-shaped Capsular Incision in Capsulorrhaphy During Surgery for Developmental Dysplasia of the Hip, Randomized Controlled Trial
Brief Title: Comparison Between Two Techniques of Capsulotomy During Capsulorrhaphy in Cases of Developmental Dysplasia of the Hip
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Thabet Hussien, Orthopedic surgery resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Capsulorrhaphy in DDH
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- U-shaped group (Active Comparator): Participants on which U shaped capsular incision will be used during capsulorrhaphy
  Interventions: Procedure: U shaped capsular incision during capsulorrhaphy
- T-shaped group (Active Comparator): Participants on which T shaped incision will be used during capsulorrhaphy
  Interventions: Procedure: T-shaped capsular incision diuring capsulorraphy

INTERVENTIONS:
Procedure: U shaped capsular incision during capsulorrhaphy — Incision of the capsule of the hip during open reduction of Developmental Dysplasia of the Hip,Incision is done with its base proximally. The transverse limb is 1 cm proximal to femoral neck base
  Other Names: U-shaped Capsulotomy
  Arms: U-shaped group
Procedure: T-shaped capsular incision diuring capsulorraphy — Incision of the capsule of the hip during open reduction of Developmental Dysplasia of the Hip done by two incisions: Vertical limb parallel to femoral neck axis and a transverse one parallel to the inguinal ligament resulting into two flabs.
  Other Names: T-shaped Capsulotomy
  Arms: T-shaped group

SUMMARY:
comparison of the outcome between using U-shaped incision and T-shaped incision for capsulorrhaphy in management of Developmental dysplasia of the hip

DETAILED DESCRIPTION:
Developmental dysplasia of the hip: Developmental dysplasia of the hip is a spectrum of abnormalities of the developing hip joint that ranges from shallowness of the acetabulum to capsular laxity and instability to frank dislocation . Developmental dysplasia of the hip is relatively common, occurring in 1 of 1000 live births.

When surgical intervention is decided, open reduction is needed to remove any obstacle that hinders hip reduction. Capsulorrhaphy is an essential step for minimizing instability of the hip after reduction The classic T-shaped capsular incision is done by two incisions: Vertical limb parallel to femoral neck axis and a transverse one parallel to the inguinal ligament resulting into two layers . Suturing them back is somewhat cumbersome after femoral head reduction. Therefore, the suggested technique utilizes a U-shaped incision to make re-suturing of the capsule easier with multiple stitches, and this study compares the outcome between using T-shaped incision and U-shaped incision for capsulorrhaphy after open reduction Femoral osteotomy or Pelvic osteotomy can be used in certain circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 1 year and younger than 4 years
* Unilateral or bilateral cases

Exclusion Criteria:

* Patients younger than 1 year and older than 4 years old
* Secondary hip dislocation ,neuromuscular disorders (as cerebral palsy, myelodysplasia or arthrogryposis).
* Patients who will undergo femoral shortening.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Modified Mackay's criteria as a clinical evaluation method | 1 year
  Postoperative clinical evaluation Grade 1(Excellent):Painless,stable hip,no limp,more than 15 degrees of internal rotation Grade 2(Good):Painless,stable hip,slight limp or decreased motion;negative trendelenburg's sign Grade 3(Fair):Minimum pain,moderate stiffness;Positive trendelenburg sign Grade 4(Poor):Significant pain

SECONDARY OUTCOMES:
Operative time ofcapsulorrhaphy | 1 year
  calculate the time needed to close the capsule of the hip
Number of stitches taken during capsulorrhaphy | 1 year
any complication detected | 1 year
  Recurrent dislocation,pain,Avascular necrosis of the hip

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McKay DW. A comparison of the innominate and the pericapsular osteotomy in the treatment of congenital dislocation of the hip. Clin Orthop Relat Res. 1974 Jan-Feb;(98):124-32. doi: 10.1097/00003086-197401000-00013. No abstract available. PMID 4817221
- [Background] Glorion C. Surgical reduction of congenital hip dislocation. Orthop Traumatol Surg Res. 2018 Feb;104(1S):S147-S157. doi: 10.1016/j.otsr.2017.04.021. Epub 2017 Dec 2. PMID 29203431
- [Background] Elbaseet HM, Abdelzaher MA. U-shaped hip capsular incision: An easier way to do hip capsulorrhaphy in developmental dysplasia of the hip - Technical note. Orthop Traumatol Surg Res. 2024 Jun;110(4):103625. doi: 10.1016/j.otsr.2023.103625. Epub 2023 Apr 21. PMID 37086945
- [Background] Zargarbashi R, Bozorgmanesh M, Panjavi B, Vosoughi F. The path to minimizing instability in developmental dysplasia of the hip: is Capsulorrhaphy a necessity or a futile habit? BMC Musculoskelet Disord. 2021 Feb 17;22(1):199. doi: 10.1186/s12891-021-04065-3. PMID 33596895
- [Background] Li Y, Hu W, Xun F, Lin X, Li J, Yuan Z, Liu Y, Canavese F, Xu H. Risk factors associated with unsatisfactory hip function in children with late-diagnosed developmental dislocation of the hip treated by open reduction. Orthop Traumatol Surg Res. 2020 Nov;106(7):1373-1381. doi: 10.1016/j.otsr.2020.03.018. Epub 2020 Jun 19. PMID 32571742
- See also: Smith's anesthesia for infants and children — https://pubs.asahq.org/anesthesiology/article/105/4/863/6744/Smith-s-Anesthesia-for-Infants-and-Children-7th
- See also: 6-Articular mobility in an African population. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1006136/
- See also: 7-persistent joint laxity and congenital dislocation of the hip — https://boneandjoint.org.uk/article/10.1302/0301-620x.46b1.40